CLINICAL TRIAL: NCT00002744
Title: Randomized Comparisons of Oral Mercaptopurine vs Oral Thioguanine and IT Methotrexate vs ITT for Standard Risk Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy in Treating Children With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1952; CCG-1952; CDR0000064665 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-09-01 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; asparaginase erwinia chrysanthemi recombinant; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Doxorubicin; Mercaptopurine; Methotrexate; pegaspargase; Prednisone; Hydrocortisone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Therapy defined in description.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy
- Arm 2 (Experimental): Therapy defined in description.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy
- Arm 3 (Experimental): Therapy defined in description.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy
- Arm 4 (Experimental): Therapy defined in description.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: therapeutic hydrocortisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: asparaginase
  Other Names: L-Asparaginase - Erwinia; NSC-106977
Drug: cyclophosphamide
  Other Names: Cytoxan; NSC-26271.
Drug: cytarabine
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar-U
Drug: daunorubicin hydrochloride
  Other Names: NSC-82151
Drug: dexamethasone
  Other Names: Decadron; NSC-34521
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC-123127
Drug: mercaptopurine
  Other Names: 6-MP; Purinethol
Drug: methotrexate
  Other Names: NSC-740
Drug: pegaspargase
  Other Names: PEG Asparaginase; Oncaspar®
Drug: prednisone
  Other Names: NSC-10023
Drug: therapeutic hydrocortisone
Drug: thioguanine
  Other Names: 6-TG; NSC-752
Drug: vincristine sulfate
  Other Names: Oncovin; NSC-67574
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways may kill more cancer cells. It is not yet known which regimen of combination chemotherapy is more effective for acute lymphoblastic leukemia

PURPOSE: Randomized phase III trial to compare different regimens of combination chemotherapy in treating children who have newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify response related factors predictive of relapse among children with previously untreated standard risk acute lymphoblastic leukemia (ALL). II. Determine the prognostic significance of residual leukemic blasts at specific times during induction therapy: M3 marrow status (greater than 25% blasts) at day 7; M2 status (5%-25% blasts) at day 14; and residual circulating leukemic blasts at days 7 and 14. III. Determine the prognostic significance of residual leukemic burden, as measured by fluorescence activated cell sorting/leukemic progenitor cell assay, on marrow aspirates acquired at the end of induction therapy, at the beginning of maintenance therapy, and at the completion of all therapy in patients with B precursor ALL. IV. Determine the prognostic significance of residual t(1;19) detected in marrow aspirates by PCR-based analyses of the fusion transcript E2A-PBX1 at the end of induction therapy, at the beginning of maintenance therapy, and at the completion of all therapy. V. Examine the interrelationships among these response-related prognostic factors and their correlation with ploidy, karyotype, and immunophenotype. VI. Determine, in a randomized study, whether substitution of oral thioguanine (TG) for oral mercaptopurine (MP) during consolidation, interim maintenance, and maintenance therapy improves event-free survival for patients with standard-risk ALL. VII. Study and compare the cellular pharmacokinetics of oral MP and oral TG during interim maintenance and maintenance therapy in selected patients. VIII. Compare the concentrations of MP and TG red blood cell metabolites (i.e., nucleotides, nucleosides, free bases, and methylated metabolites) during interim maintenance and maintenance therapy, and determine whether low levels of metabolites predict relapse in selected patients. IX. Determine the activities of thiopurine methyltransferase and hypoxanthine guanine phosphoribosyl transferase several times during interim maintenance and maintenance treatment, and compare the activities between the two thiopurine treatment groups in selected patients. X. Compare the incidence of central nervous system (CNS) relapse and event-free survival in patients receiving intrathecal methotrexate (MTX) vs. triple intrathecal chemotherapy (MTX/cytarabine/hydrocortisone) for presymptomatic CNS treatment. XI. Determine whether cerebrospinal fluid (CSF) terminal deoxynucleotidyl transferase (TdT) positivity predicts for CNS or marrow relapse by measuring TdT activity on CSF cytospins in cases with low white blood cell count (less than 5 cells per cubic millimeter) and suspected or questionable "blasts" during maintenance therapy. XII. Determine event-free survival in patients with standard-risk ALL and M3 marrow at day 14 when treated with intensive therapy designed for higher-risk ALL.

OUTLINE: This is a randomized study. Patients are stratified according to participating institution. The following acronyms are used: ARA-C Cytarabine, NSC-63878 ASP Asparaginase (E. coli), NSC-109229 CTX Cyclophosphamide, NSC-26271 DM Dexamethasone, NSC-34521 DNR Daunorubicin, NSC-82151 DOX Doxorubicin, NSC-123127 HC Hydrocortisone, NSC-10483 MP Mercaptopurine, NSC-755 MTX Methotrexate, NSC-740 PEG-ASP Pegaspargase, NSC-624239 PRED Prednisone, NSC-10023 TG Thioguanine, NSC-752 TIT Triple Intrathecal Therapy (IT MTX/IT ARA-C/IT HC) VCR Vincristine, NSC-67574 Induction: All patients receive oral PRED on days 0-27, VCR IV on days 0, 7, 14, and 21, and ASP IM 3 times a week for 3 weeks beginning on day 2-4. ARA-C IT is administered on day 0, and MTX IT is administered on days 7 and 28 (days 7, 14, 21, and 28 if CNS disease at diagnosis). Following Induction, patients who achieve remission are randomly assigned to 1 of 4 treatment arms. Arm I: Consolidation (begins day 28 of Induction): PRED is tapered from Induction over 10 days. Patients receive VCR IV on day 0, oral MP on days 1-27, and MTX IT on days 7, 14, and 21 (only day 7 if CNS disease at diagnosis). Interim Maintenance 1 (begins day 28 of Consolidation): Patients receive oral PRED on days 0-4 and 28-32, VCR IV days 0 and 28, oral MTX on days 0, 7, 14, 21, 28, 35, 42, and 49, and oral MP on days 0-49. Delayed Intensification 1 (begins day 56 of Interim Maintenance 1): Patients receive oral DM on days 0-6 and 14-20, VCR IV on days 0, 7, and 14, DOX IV over 15-120 min on days 0, 7, and 14, ASP IM twice a week for 2 weeks beginning day 2-4, CTX IV over 20-30 min on day 28, oral TG on days 28-41, ARA-C IV or SC on days 29-32 and 36-39, and MTX IT on days 0, 28, and 35. Interim Maintenance 2 (begins day 56 of Delayed Intensification 1): Patients receive PRED/VCR/MTX/MP as in Interim Maintenance 1. Delayed Intensification 2 (begins day 56 of Interim Maintenance 2): Patients receive DM/VCR/DOX/ASP, CTX/TG/ARA-C, and MTX IT as in Delayed Intensification 1. Maintenance (begins day 56 of Delayed Intensification 2): Patients receive oral PRED on days 0-4, 28-32, and 56-60, VCR IV on days 0, 28, and 56, oral MP on days 0-83, oral MTX on days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, and 77 (omitted during wk of IT therapy), and MTX IT on day 0. Treatment continues every 84 days for 2 years (girls) or 3 years (boys) from the beginning of Interim Maintenance 1. Arm II: Patients receive treatment as in arm I, except TIT is TIT substituted for MTX IT. Arm III: Patients receive treatment as in arm I with oral TG substituted for oral MTX in Consolidation, Interim Maintenance 1 and 2, and Maintenance. If secondary veno-occlusive disease occurs, MP is substituted for TG during Maintenance. Arm IV: Patients receive treatment as in arm III with TIT substituted for MTX IT. If secondary veno-occlusive disease occurs, MP is substituted for TG during Maintenance. Patients with M3 marrow after 2 weeks or M2 marrow after 4 weeks of Induction, or with Philadelphia chromosome (t[9;22][q34;q11]), t(4;11)(q21;q23), or hypodiploidy, proceed to the following more intensive treatment regimen for further therapy: Induction (begins day 14 to day 19 of initial Induction): Patients receive oral PRED on days 14-27, VCR IV on days 14 and 21 (day 14 dose omitted if day 14 dose from original Induction already given), DNR IV continuously on days 14-16 (48 hours total), ASP IM three times a week for 9 total doses (including those received on original Induction), MTX IT on days 28 and 35 (days 21, 28, and 35 if CNS disease at diagnosis). Patients with M1/M2 bone marrow after day 35 proceed to Consolidation. Consolidation (begins day 28 or 35 of Induction in this regimen, depending on timing of entry on this regimen): PRED is tapered from Induction over 10 days. Patients receive CTX IV 20-30 minutes on days 0 and 28, oral MP on days 0-13 and 28-41, ARA-C IV or SC on days 1-4, 8-11, 29-32, and 36-39, VCR IV on days 14, 21, 42, and 49, PEG-ASP IM on days 14 and 42, and MTX IT on days 7, 14, and 21 (only day 7 if CNS disease at diagnosis). Patients with M1 or M2 marrow and no extramedullary leukemia after day 63 proceed to Interim Maintenance 1. Interim Maintenance 1 (begins day 63 of Consolidation): Patients receive VCR IV on days 0, 10, 20, 30, and 40, MTX IV on days 0, 10, 20, 30, and 40, and PEG-ASP IM on days 1 and 21. Patients with M1 bone marrow after day 56 proceed to Delayed Intensification I. Delayed Intensification 1 (begins day 56 of Interim Maintenance 1): Patients receive oral DM on days 0-6 and 14-20, VCR IV on days 0, 7, 14, 42, and 49, DOX IV over 15-120 minutes on days 0, 7, and 14, PEG-ASP IM on days 3 and 42, CTX IV over 20-30 minutes on day 28, oral TG on days 28-41, ARA-C IV or SC on days 29-32 and 36-39, and MTX IT on days 28 and 35. Interim Maintenance 2 (begins day 56 of Delayed Intensification 1): Patients receive VCR/MTX/PEG-ASP as in Interim Maintenance 1, and MTX IT on days 0, 20, and 40. Delayed Intensification 2 (begins day 56 of Interim Maintenance 2): Patients receive DM/VCR/DOX/PEG-ASP, CTX/TG/ARA-C, and MTX IT as in Delayed Intensification 1. Maintenance (begins day 56 of Delayed Intensification 2): Patients receive PRED/VCR/MP/MTX, and MTX IT as in arm I Maintenance. Patients with CNS or testicular involvement at diagnosis receive appropriate radiotherapy concurrent with Consolidation. Radiotherapy begins within 4 days of initiation of Consolidation. Craniospinal irradiation is given 5 days a week. Testicular irradiation is given to both testes 5 days a week over 2-3 weeks. Patients are followed every 6-8 weeks during year 1, every 3 months during year 2, every 6 months during year 3, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1970 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed acute lymphoblastic leukemia (ALL) obtained by bone marrow aspirate or bone marrow biopsy No greater than 25% L3 blasts Initial white blood cell count less than 50,000/mm3 (performed at CCG institution) Massive lymphadenopathy, massive splenomegaly, and/or large mediastinal mass allowed CNS or testicular leukemia allowed Allogeneic bone marrow transplant should be considered (if donor available) for patients with Philadelphia chromosome (t[9;22][q34;q11]) or translocation (4;11)(q21;q23)

PATIENT CHARACTERISTICS: Age: 1 through 9 Performance status: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: No prior treatment for ALL Biologic therapy: Not specified Chemotherapy: Intrathecal cytarabine (IT ARA-C) may begin prior to registration provided systemic chemotherapy initiated within 72 hours after IT ARA-C Endocrine therapy: See Radiotherapy At least 1 month since prior systemic steroids Steroids given for less than 48 hours allowed Inhaled corticosteroids allowed at any time Radiotherapy: Radiotherapy or dexamethasone for mediastinal mass causing superior mediastinal syndrome allowed prior to registration, if indicated Surgery: Not specified

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1970 (Actual)
Dates: Start 1996-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival
  Primary outcome index used in examining the randomized treatment groups will be event-free survival (EFS) from the time of randomization (i.e., end of Induction), where the life table events will consist of the first occurrence of leukemic relapse at any site, death, or occurrence of a second malignancy.

SECONDARY OUTCOMES:
Comparisons of CNS relapse incidence rates
  Comparisons of CNS relapse incidence rates for the IT MTX versus ITT groups is also planned as an important endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Linda C. Stork, MD, Study Chair — Doernbecher Children's Hospital at Oregon Health and Science University
Locations (34):
- United States (31):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Background] Matloub Y, Asselin BL, Stork LC, et al.: Outcome of children with T-Cell acute lymphoblastic leukemia (T-ALL) and standard risk (SR) features: results of CCG-1952, CCG-1991 and POG 9404. [Abstract] Blood 104 (11): A-680, 195a, 2004.
- [Result] Stork LC, Matloub Y, Broxson E, La M, Yanofsky R, Sather H, Hutchinson R, Heerema NA, Sorrell AD, Masterson M, Bleyer A, Gaynon PS. Oral 6-mercaptopurine versus oral 6-thioguanine and veno-occlusive disease in children with standard-risk acute lymphoblastic leukemia: report of the Children's Oncology Group CCG-1952 clinical trial. Blood. 2010 Apr 8;115(14):2740-8. doi: 10.1182/blood-2009-07-230656. Epub 2010 Feb 1. PMID 20124218
- [Result] Kadan-Lottick NS, Brouwers P, Breiger D, Kaleita T, Dziura J, Northrup V, Chen L, Nicoletti M, Bostrom B, Stork L, Neglia JP. Comparison of neurocognitive functioning in children previously randomly assigned to intrathecal methotrexate compared with triple intrathecal therapy for the treatment of childhood acute lymphoblastic leukemia. J Clin Oncol. 2009 Dec 10;27(35):5986-92. doi: 10.1200/JCO.2009.23.5408. Epub 2009 Nov 2. PMID 19884541
- [Result] Malempati S, Gaynon PS, Sather H, La MK, Stork LC; Children's Oncology Group. Outcome after relapse among children with standard-risk acute lymphoblastic leukemia: Children's Oncology Group study CCG-1952. J Clin Oncol. 2007 Dec 20;25(36):5800-7. doi: 10.1200/JCO.2007.10.7508. PMID 18089878
- [Result] Matloub Y, Lindemulder S, Gaynon PS, Sather H, La M, Broxson E, Yanofsky R, Hutchinson R, Heerema NA, Nachman J, Blake M, Wells LM, Sorrell AD, Masterson M, Kelleher JF, Stork LC; Children's Oncology Group. Intrathecal triple therapy decreases central nervous system relapse but fails to improve event-free survival when compared with intrathecal methotrexate: results of the Children's Cancer Group (CCG) 1952 study for standard-risk acute lymphoblastic leukemia, reported by the Children's Oncology Group. Blood. 2006 Aug 15;108(4):1165-73. doi: 10.1182/blood-2005-12-011809. Epub 2006 Apr 11. PMID 16609069
- [Result] Bassal M, La MK, Whitlock JA, Sather HN, Heerema NA, Gaynon PS, Stork LC. Lymphoblast biology and outcome among children with Down syndrome and ALL treated on CCG-1952. Pediatr Blood Cancer. 2005 Jan;44(1):21-8. doi: 10.1002/pbc.20193. PMID 15368546
- [Result] Malempati S, Gaynon PS, Sather H, et al.: Outcome after relapse among children with standard risk (SR) ALL treated on CCG-1952. [Abstract] Blood 104 (11): A-520, 2004.
- [Result] Stork LC, Sather H, Hutchinson RJ, et al.: Comparison of mercaptopurine (MP) with thioguanine (TG) and IT methotrexate (ITM) with IT "triples" (ITT) in children with SR-ALL: results of CCG-1952. [Abstract] Blood 100 (11 Pt 1): A-585, 156a, 2002.
- [Result] Stork LC, Sather H, Yanofsky R, et al.: Hyperdiploidy with trisomy 10 and TEL-AML1 expression among children with standard risk acute lymphoblastic leukemia (SR-ALL): a CCG-1952 report. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1476, 2001.
- [Result] Gaynon PS, Stork L, Sather H, et al.: Leukemic progenitor cell content of pre- and post-induction chemotherapy bone marrow specimens from children with newly diagnosed or relapsed acute lymphoblastic leukemia (ALL). [Abstract] Proceedings of the American Society of Clinical Oncology 18: A-2187, 567a, 1999.
- [Result] Stork LC, Erdmann G, Adamson P, et al.: Oral 6-thioguanine causes relatively mild and reversible hepatic veno-occlusive disease(VOD). J Pediatr Hematol Oncol 20: 400a, 1998.